CLINICAL TRIAL: NCT01345864
Title: A Randomized, Double-Blind, Sponsor Unblinded, Placebo- And Positive- Controlled Study To Evaluate The Effects Of Single Oral Administrations Of PF-04995274, Alone Or In Combination With Donepezil, On Scopolamine-Induced Deficits In Psychomotor And Cognitive Function In Healthy Adults
Brief Title: Assessment Of The Effects Of Single Doses Of An Investigational Drug, Given Alone Or With Donepezil, On Scopolamine-Induced Changes In Memory And Learning In Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B1661006
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: attention cognition memory problem solving scopolamine challenge
MeSH Terms: interventions — Scopolamine; Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort A (Other): Parallel design with 5 unique treatment groups Donepezil tablets and matching placebo tablets may be overencapsulated as needed.
  Interventions: Drug: Scopolamine + Donepezil Placebo + PF-04995274 Placebo; Drug: Scopolamine + Donepezil 5 mg + PF-04995274 Placebo; Drug: Scopolamine + Donepezil 10mg + PF-04995274 Placebo; Drug: Scopolamine + Donepezil Placebo + PF-04995274 0.25 mg; Drug: Scopolamine + Donepezil Placebo + PF-04995274 15 mg

INTERVENTIONS:
Drug: Scopolamine + Donepezil Placebo + PF-04995274 Placebo — Scopolamine 0.5 mg subcutaneously x 1 dose on Day 1 Donepezil-matching placebo tablet x 1 dose on Day 1 PF-04995274 matching placebo oral liquid x 1 dose on Day 1
Drug: Scopolamine + Donepezil 5 mg + PF-04995274 Placebo — Scopolamine 0.5 mg subcutaneously x 1 dose on Day 1 Donepezil 5 mg tablet orally x 1 dose on Day 1 PF-04995274 matching placebo oral liquid x 1 dose on Day 1
Drug: Scopolamine + Donepezil 10mg + PF-04995274 Placebo — Scopolamine 0.5 mg subcutaneously x 1 dose on Day 1 Donepezil 10 mg (2 x 5 mg tablets) orally x 1 dose on Day 1 PF-04995274 matching placebo oral liquid x 1 dose on Day 1
Drug: Scopolamine + Donepezil Placebo + PF-04995274 0.25 mg — Scopolamine 0.5 mg subcutaneously x 1 dose on Day 1 Donepezil-matching placebo tablet x 1 dose on Day 1 PF-04995274 0.25 mg oral liquid x 1 dose on Day 1
Drug: Scopolamine + Donepezil Placebo + PF-04995274 15 mg — Scopolamine 0.5 mg subcutaneously x 1 dose on Day 1 Donepezil-matching placebo tablet x 1 dose on Day 1 PF-04995274 15 mg oral liquid x 1 dose on day 1

SUMMARY:
This study is designed to look at the potential for an investigational drug (PF-04995274, under development by Pfizer, Inc. as a potential treatment for Alzheimer's disease) to reverse changes in memory and learning/problem solving skills caused by co-administration of a marketed drug called scopolamine. Scopolamine is known to cause temporary changes in memory and learning/problem solving skills that are similar to those seen in people with alzheimer's disease(AD).

DETAILED DESCRIPTION:
Changes in sponsor's organizational strategy have led to the decision to terminate the study and therefore to not conduct the second cohort (Cohort B/arms 2 and 3) . This decision was not based on significant safety concerns. Date of termination (ie, the date the site was notified to stop study activities) was 12 Oct 2011.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers; females must be of non-childbearing potential.
* Weight with normal limits for height.
* Willing to comply with study schedule and able to complete 2 practice sessions (pre-study) with computerized memory and learning/problem solving tests.

Exclusion Criteria:

* Positive urine drug screen; concurrent use of prescription or over-the-counter (OTC) drugs or dietary supplements within 7 days or 5 half-lives prior to the first dose of study medication.
* Use of medications with significant serotonergic, cholinergic or anticholinergic side effects [SSRIs, pyridostigmine, tricyclic antidepressants, meclizine, oxybutynin]) within 4 weeks of first dose of study drug.
* Glaucoma
* Abnormal electrocardiogram (ECG)
* Treatment with an investigational drug within 30 days of dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Groton Maze Learning Test (Total Errors) | Day 1 of each period at 8 time points from 0-12 hr postdose relative to scopolamine dosing

SECONDARY OUTCOMES:
Detection Task (Speed; included in CogState test battery) | Day 1 of each period at 8 time points from 0-12 hrs postdose relative to scopolamine dosing
Identification Task (Speed; included in CogState test battery) | Day of each period at 8 time points from 0-12 hrs postdose relative to scopolamine dosing
One Card Learning Task (Accuracy of Performance; included in CogState test battery) | Day 1 of each period at 8 time points from 1-12 hrs postdose relative to scopolamine dosing
Bond-Lader Visual Analogue Scales | Day 1 of each period at 8 time points from 1-12 hours postdose relative to scopolamine dosing

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1661006&StudyName=Assessment%20Of%20The%20Effects%20Of%20Single%20Doses%20Of%20An%20Investigational%20Drug%2C%20Given%20Alone%20Or%20With%20Donepezil%2C%20On%20Scopolamine-Induced%20Changes%20